CLINICAL TRIAL: NCT04334252
Title: Descriptive Study Regarding the Ambulant Screening Protocol for COVID-19 in Times of High SARS CoV-2 Prevalence
Brief Title: Descriptive Study Regarding Ambulant Screening During COVID-19 Pandemia
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Ina Callebaut, dr, Jessa Hospital
Other Study IDs: JessaH_COVID19_prescreening
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
Descriptive prospective study to investigate the prevalence of COVID 19 during ambulant screening

DETAILED DESCRIPTION:
The exact prevalence of COVID-19 is unknown. Due to the relatively high number of diagnosed, symptomatic infections despite a strict policy, we expect a high prevalence of COVID 19 throughout the entire population. The risk that an asymptomatic carrier who is admitted to the hospital for a (semi)urgent surgery, treatment of investigation transfers the virus to the hospital staff is very high, and vice versa. This risk is even higher during surgery, where intubation is necessary. Therefore we would like to pre-screen all patients ambulantly on the presence of COVID 19 since there is no consensus for screening at the moment. The golden standard is the SARS CoV-2 PCR on the nasopharyngeal sample together with a CT scan of the lungs. Patients in which a bloodsample is taken as standard of care procedure in this ambulant screening will be asked to give more blood for further investigation.

On top of this standard of care screening, we will perform a questionnaire at the pre-operative visit which evaluates the possible occurence of certain symptoms in the last 2 weeks. These symptoms are fever, anorexia, cough, diarrhea, sneezing, vomiting, dyspnea, headache, rhinorrhea, loss of smell, muscle pain, sputum, sore throat and fatigue. Patients were also asked if one of their housemates are affected by these symptoms. Furthermore, 2 weeks after surgery, patient will be contacted to phone in order to fill the same questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > 18 years scheduled for a (semi) urgent surgery, hematological or oncological treatment or elektrophysiciological investigations in the Jessa hospital

Exclusion Criteria:

* Patients < 18 years
* Adult patients who are unable the give informed consent
* Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients scheduled for a (semi) urgent surgery, hematological or oncological treatment or elektrophysiciological investigations in the Jessa hospital and seen at the pre-operative consultation will be asked to participate and to fullfill the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 528 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of symptoms | at the ambulant screening
  Prevalence of fever, cough, anorexia, fatigue, diarrhea, vomiting, dyspnee, sore throat and sputum
Prevalence of positive Sars CoV-2 PCR | at the ambulant screening
  Prevalence of positive COVID 19 tests in patients planned for surgery, treatment or investigation in the hospital
Prevalence of positive radiological findings | at the ambulant screening
  Prevalence of positive radiological findings in CT scans of the lungs of planned for surgery, treatment or investigation in the hospital

SECONDARY OUTCOMES:
Prediction of symptoms | 2 weeks after surgery or treatment
  Prediction of symptoms of COVID 19, based on evaluated baseline questionnaire
Prediction of symptoms | 2 weeks after surgery or treatment
  Prediction of symptoms of COVID 19, based on radiological findings of CT scans
Prediction of symptoms | 2 weeks after surgery or treatment
  Prediction of symptoms of COVID 19, based on COVID 19 PCR results

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No